CLINICAL TRIAL: NCT05150938
Title: Observational Studies in Cancer Associated Thrombosis for Rivaroxaban in SwEden (OSCAR-SE)
Brief Title: A Study to Gather Information About Rivaroxaban in Patients in Sweden With Cancer Who Also Have Thrombosis (OSCAR-SE)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 21616
Record Dates: First submitted 2021-11-18; First posted 2021-12-09 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Treatment of Venous Thromboembolism in Cancer Patients
MeSH Terms: interventions — Rivaroxaban; Heparin, Low-Molecular-Weight; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients with VTE: Cancer patients who received anticoagulation treatment.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Low molecular weight heparin (LMWH); Drug: vitamin K antagonist (VKA); Drug: other NOACs

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Retrospective cohort analysis using Swedish registries including the Cancer Registry, National Patient Registry, Prescribed Drug Registry, and Cause of Death Registry.
Drug: Low molecular weight heparin (LMWH) — Retrospective cohort analysis using Swedish registries including the Cancer Registry, National Patient Registry, Prescribed Drug Registry, and Cause of Death Registry.
Drug: vitamin K antagonist (VKA) — Retrospective cohort analysis using Swedish registries including the Cancer Registry, National Patient Registry, Prescribed Drug Registry, and Cause of Death Registry.
Drug: other NOACs — Retrospective cohort analysis using Swedish registries including the Cancer Registry, National Patient Registry, Prescribed Drug Registry, and Cause of Death Registry.

SUMMARY:
This is an observational study in which patient data from the past on venous thromboembolism (VTE) in patients with cancer is studied.

VTE is a condition in which a patient has problems due to the formation of blood clots in the veins. Blood clots can reduce the flow of blood to vital organs such as the heart and lungs, which can lead to them becoming damaged. VTE can also be "recurrent". This means that the blood clots have returned after treatment. People who have cancer have an increased risk of developing VTE.

Three main types of anticoagulation treatments ("blood thinners") have been available for patients with cancer who also have VTE

* Low molecular weight heparins (LMWHs)
* Vitamin K antagonists (VKAs)
* Non-vitamin K antagonist oral anticoagulants (NOACs) The treatment rivaroxaban belongs to the NOACs.

Compared to other treatments available to patients who have cancer and VTE, NOACs may cause fewer medical problems and can be easier for patients to take correctly.

In this study, the researchers will collect data about:

* the type of VTE treatments given and for how long the treatments are taken
* the risk of blood clots returning in the veins after treatment, any events of major bleeding, and the number of deaths in patients with cancer who do not have a high risk of bleeding

The researchers will compare this information in the patients

* who received rivaroxaban to the patients who received LMWHs
* who received NOACs to the patients who received LMWHs.

There will be no required visits with a study doctor or required tests in this study. The researchers will look at the health information from adult patients in Sweden who were diagnosed with cancer between 2013 and 2019 and also have VTE. The researchers will collect this information from Swedish health registers including the Cancer Registry, National Patient Registry, Prescribed Drug Registry, and Cause of Death Registry.

ELIGIBILITY:
Inclusion Criteria:

* A resident in Sweden of 18+ years of age
* A Swedish Person Identification Number
* A diagnosis of cancer ((ICD10 = C00-C97) in the Swedish Cancer registry during 2013-2019 and a diagnosis of VTE subsequent to the cancer diagnosis.

Exclusion Criteria:

* A diagnosis of atrial fibrillation, total hip or knee replacement or acute coronary syndrome (for evaluation of treatment patterns) before the date of VTE diagnosis
* A dispensed prescription for any oral anticoagulant (OAC) before the date of VTE diagnosis
* A cancer diagnosis associated with high bleeding risk, including upper gastrointestinal cancer, malignant immunoproliferative diseases and leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with cancer in Sweden from year 2013 to 2019.
Sampling Method: Non-Probability Sample
Enrollment: 5737 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Recurrence of VTE | Retrospective data analysis from 2013 to 2020
Major bleedings | Retrospective data analysis from 2013 to 2020
All-cause death | Retrospective data analysis from 2013 to 2020
Choice of anticoagulation treatments for VTE | Retrospective data analysis from 2013 to 2020
Duration of anticoagulation treatments for VTE | Retrospective data analysis from 2013 to 2020
Recurrence of VTE with different treatment types of LMWH, VKA and NOAC | Retrospective data analysis from 2013 to 2020
Major bleedings with different treatment types of LMWH, VKA and NOAC | Retrospective data analysis from 2013 to 2020
All-cause death with different treatment types of LMWH, VKA and NOAC | Retrospective data analysis from 2013 to 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish registries, Multiple Locations, Many Locations, Sweden

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Linder M, Ekbom A, Brobert G, Vogtlander K, Balabanova Y, Becattini C, Carrier M, Cohen AT, Coleman CI, Khorana AA, Lee AYY, Psaroudakis G, Abdelgawwad K, Rivera M, Schaefer B, Giunta DH. Comparison of rivaroxaban and low molecular weight heparin in the treatment of cancer-associated venous thromboembolism: a Swedish national population-based register study. J Thromb Thrombolysis. 2024 Aug;57(6):973-983. doi: 10.1007/s11239-024-02992-1. Epub 2024 May 12. PMID 38735015